CLINICAL TRIAL: NCT06189404
Title: A Phase 1, Open-Label, Drug-Drug Interaction Study to Evaluate the Effect of Multiple Oral Doses of Tigulixostat on the Pharmacokinetics of a Single Oral Dose of Theophylline
Brief Title: Effect of Tigulixostat on the Pharmacokinetics of Theophylline
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: LG Chem (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: LG-GDCL013
Record Dates: First submitted 2023-12-07; First posted 2024-01-03 (Actual); Last update posted 2024-01-03 (Actual); Status verified 2023-12

CONDITIONS: Gout; Hyperuricemia
MeSH Terms: conditions — Gout; Hyperuricemia | interventions — Theophylline

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Cohort 1 (Periods 1-3), Cohort 2 (Periods 1-4) (Experimental): Period 1: Single oral dose of theophylline (Day 1); Period 2: Once-daily oral doses of tigulixostat (Days 6 to 10); Period 3: Once-daily oral doses of tigulixostat (Days 11 to 13) and a single oral dose of theophylline (Day 11); Period 4: Single oral dose of tigulixostat (Day 19)
  Interventions: Drug: Tigulixostat; Drug: Theophylline

INTERVENTIONS:
Drug: Tigulixostat — 300 mg oral dose
  Other Names: LC350189
Drug: Theophylline — 400 mg oral dose

SUMMARY:
A phase 1, open-label, drug-drug interaction study to evaluate the effect of multiple doses of tigulixostat on the pharmacokinetics of single-dose theophylline in healthy adult volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, Ages 18 to 55, inclusive.
* BMI 18.0 - 32.0 kg/m2, inclusive, at screening.
* In good general health as determined by medical history, clinical laboratory assessments, vital sign measurements, 12-lead ECG results, and physical examination findings at screening.
* Females of childbearing potential and males who agree to use contraception. Non-pregnant, non-lactating females who must have a negative pregnancy test at screening and check-in.

Exclusion Criteria:

* Significant history or indications of ill-health, as judged by the investigator.
* Any surgical or medical condition(s) possibly affecting drug absorption, distribution, metabolism, and excretion.
* eGFRcr of <60 (mL/min)/1.73 m2 at screening.
* alanine aminotransferase, aspartate aminotransferase, or total bilirubin ≥2 times the upper limit of normal at screening and check-in.
* Used any prescription or over-the-counter medications (except acetaminophen [Tylenol] up to 2 g per day), including herbal or nutritional supplements, within 14 days before the first dose of study drug.
* Consumed grapefruit or grapefruit juice, Seville orange or Seville orange-containing products (eg, marmalade), or caffeine- or xanthine-containing products within 48 hours before the first dose of study drug.
* History of hypersensitivity to theophylline or other xanthines and tigulixostat.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2023-10-31 (Actual); Primary Completion 2023-11-13 (Actual); Study Completion 2023-11-30 (Actual)

PRIMARY OUTCOMES:
AUC0-t of theophylline with and without tigulixostat | Up to 72 hours
AUC0-inf of theophylline with and without tigulixostat | Up to 72 hours
Cmax of theophylline with and without tigulixostat | Up to 72 hours

SECONDARY OUTCOMES:
Incidence of reported adverse events (AEs) | Up to Day 28
AUC0-t of tigulixostat and metabolite GD-MET-1 | Up to 24 hours
Cmax of tigulixostat and metabolite GD-MET-1 | Up to 24 hours

CONTACTS AND LOCATIONS:
Locations (1):
- PPD - Austin Research Unit, Austin, Texas, United States